CLINICAL TRIAL: NCT02326883
Title: UH3 Pragmatic Trial of Population-based Programs to Prevent Suicide Attempt
Brief Title: UH3 Pragmatic Suicide Prevention Trial
Acronym: SPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); HealthPartners Institute (Other); National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4UH3MH007755 (NIH); UH2AT007755 (NIH); UH3MH007755 (NIH)
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Depression; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Care Management (Experimental): The Care Management intervention will last up to a year and includes routine outreach to assess ongoing risk of suicide attempt, and care management to monitor and facilitate ongoing engagement in outpatient follow-up. The Care Manager will coordinate care with treating mental health and primary care providers (ongoing usual care) using Epic Staff Messaging (or telephone contacts if necessary).
  Interventions: Behavioral: Care Management
- Skills Training (Experimental): The Skills Training intervention will last up to a year and uses an online skills training program to support patients in developing and using self-management skills for emotion regulation and crisis management. A Coach will monitor each participant's use of the program and send periodic messages (using Epic secure messaging) to encourage and support use of the program and practice of program skills.
  Interventions: Behavioral: Skills Training
- Usual Care (Active Comparator): Those assigned to the Usual Care group will not be approached or contacted.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Care Management — The Care Management intervention includes routine outreach to assess ongoing risk of suicide attempt and care management to monitor and facilitate ongoing engagement in outpatient follow-up. The Care Manager will coordinate care with treating mental health and primary care providers (ongoing usual care) using Epic Staff Messaging (or telephone contacts if necessary).
  Arms: Care Management
Behavioral: Skills Training — The Skills Training intervention uses an online skills training program to support patients in developing and using self-management skills for emotion regulation and crisis management. A Coach will monitor each participant's use of the program and send periodic messages (using Epic secure messaging) to encourage and support use of the program and practice of program skills.
  Arms: Skills Training
Behavioral: Usual Care — Those assigned to usual care will not be contacted at all by study staff and will continue to receive usual care from treating primary care and mental health providers.
  Arms: Usual Care

SUMMARY:
This pragmatic clinical trial will evaluate the effectiveness of two population-based outreach programs for preventing suicide attempts among patients identified as at-risk. The study will be conducted at Kaiser Permanente (KP) Washington (the lead site) and at HealthPartners, KP Colorado and KP Northwest. Electronic health records will be used to identify outpatients aged 18 or older who respond to a routinely administered PHQ depression questionnaire by reporting thoughts of death or self-harm "most of the days" or "nearly every day". This trial will be limited to patients receiving care from one of the four participating health systems. Eligible patients will be automatically assigned to continue in usual care (1/3) or to either of the two intervention programs (1/3 each). Those assigned to usual care will not be contacted at all by study staff and will continue to receive usual care from treating primary care and mental health providers. Both intervention programs involve outreach by Epic secure messaging (with optional telephone outreach for those not reading messages). The Care Management intervention includes routine outreach to assess ongoing risk of suicide attempt and care management to monitor and facilitate ongoing engagement in outpatient follow-up. The Care Manager will coordinate care with treatment by primary and behavioral health care providers using Epic Staff Messaging (or telephone contacts if necessary). The Skills Training intervention uses an online skills training program to support patients in developing and using self-management skills for emotion regulation and crisis management. A Coach will monitor each participant's use of the program and send periodic messages (using Epic secure messaging) to encourage and support use of the program and practice of program skills. Each intervention continues for up to one year. In all three groups (Usual Care, Care Management, and Skills Training) virtual data warehouse data will be used to identify likely suicide attempts over 18 months following randomization. Analyses will compare risk of suicide attempt among all those randomized, regardless of response to the initial invitation or level of participation in the intervention programs. Comparison of all those randomized is the only scientifically valid method for assessing the overall impact of either program on population-level risk of suicide attempt.

DETAILED DESCRIPTION:
Each week, a programmer will use Epic/Clarity data to identify adult outpatients who completed a PHQ depression questionnaire in the previous week and reported thoughts of death or self-harm "most of the days" or "nearly every day". This trial will be limited to patients receiving care from one of the three participating health systems.

Those identified will be automatically assigned to continued Usual Care or to one of two intervention programs (Care Management or Skills Training).

The Care Management intervention includes periodic outreach to assess ongoing risk of suicide attempt and as-needed care management to facilitate engagement in ongoing outpatient follow-up. Contacts will occur by secure messaging (with the option of telephone outreach for those who do not read messages). Each contact will include a request to complete a new risk assessment questionnaire (the abbreviated Columbia Suicide Severity Rating Scale used at each site) unless a risk assessment was recently documented in the medical record. Using an algorithm tested in pilot studies, the Care Manager will determine appropriate timing of follow-up and (if not already scheduled) communicate with the participant to facilitate appropriate follow-up care. Time between outreach contacts will vary from 2 weeks to 2 months, depending on the most recent risk assessment. Outreach contacts will continue up to 12 months. All outreach contacts will be documented in the Epic electronic health record in the same manner as any other mental health clinical contacts. The Care Manager(s) will be licensed mental health clinician(s) with experience in suicide risk assessment, supervised by site specific clinician investigators. A detailed protocol for the Care Management program (including sample messages) is included with this application.

The Skills Training intervention is an online program intended to teach specific skills for emotion regulation and crisis management. The content of the program is derived from Dialectical Behavior Therapy, an evidence-based psychotherapy designed for people at risk for suicide attempts. The program includes four modules or chapters, each focused on a specific skill. Each chapter includes written and video didactic instruction, video examples, in-vivo practice, and written homework exercises. The program will be supported by a Coach who will send periodic messages (via Epic secure messaging) encouraging use of the program and practice of specific skills. Coaching messages will be scheduled every 1-3 weeks during the first 3 months of the program and every 1-3 months over the following 9 months (varying according to each participant's level of participation and progress in the program). All coaching messages will be documented in the Epic electronic health record in the same manner as any other mental health clinical contacts. The Coach(es) will be licensed mental health clinician(s) supervised by site specific clinician investigators. The online program will be delivered by a secure website (KP Washington Health Research Institute's DatStat server), and participants will reach the program using encrypted personalized links sent to them via Epic secure messaging. This trial does not have open enrollment, please see the public facing website at www.NowMattersNow.org

Those assigned to Usual Care will not be contacted.

For all patients in all three intervention groups, a site programmer will extract data from the Virtual Data Warehouse to identify probable suicide attempts over 18 months following randomization.

ELIGIBILITY:
Inclusion Criteria:

We propose to include all patients at the participating sites who:

* Complete PHQ questionnaire and respond to item 9 (regarding thoughts of death or self-harm) "more than half the days" or "nearly every day"
* Are currently enrolled in one of the four participating health systems
* Are age 18 or older
* Recent use of Epic Secure Messaging

Exclusion Criteria:

* Recorded diagnosis of dementia or developmental delay
* Previously invited to participate in the UH2 pilot trial
* Non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18882 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Simon, MD, MPH, Principal Investigator — KP Washington

IPD SHARING:
Plan to Share IPD: Yes
This person-level dataset will include the following variables:
  * Time to suicide attempt or death
  * Time to censoring for disenrollment or death from other cause
  * Age group
  * Sex
  * Race/ethnicity
  * Site of care (mental health specialty, primary care, other)
  * PHQ9 item 9 score at baseline
  * Year of enrollment
  * Intervention assignment (Skills Training, Risk Assessment/Care Management, Usual Care) We do not propose to include study site (health system) in this publicly available dataset given concerns by participating health systems that such data could be used for inappropriate comparisons of suicide attempt rates across health systems.
Supporting Information: Study Protocol, SAP
Time Frame: . Data will be available no later than publication date of primary study findings.
Access Criteria: Datasets for primary analyses will be freely shared with any interested researcher or member of the public using an unsupervised public data archive model.

REFERENCES:
- [Background] Simon GE, Beck A, Rossom R, Richards J, Kirlin B, King D, Shulman L, Ludman EJ, Penfold R, Shortreed SM, Whiteside U. Population-based outreach versus care as usual to prevent suicide attempt: study protocol for a randomized controlled trial. Trials. 2016 Sep 15;17(1):452. doi: 10.1186/s13063-016-1566-z. PMID 27634417
- [Derived] Simon GE, Shortreed SM, Rossom RC, Beck A, Clarke GN, Whiteside U, Richards JE, Penfold RB, Boggs JM, Smith J. Effect of Offering Care Management or Online Dialectical Behavior Therapy Skills Training vs Usual Care on Self-harm Among Adult Outpatients With Suicidal Ideation: A Randomized Clinical Trial. JAMA. 2022 Feb 15;327(7):630-638. doi: 10.1001/jama.2022.0423. PMID 35166800
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Whiteside U, Richards J, Simon GE. Brief Interventions via Electronic Health Record Messaging for Population-Based Suicide Prevention: Mixed Methods Pilot Study. JMIR Form Res. 2021 Apr 12;5(4):e21127. doi: 10.2196/21127. PMID 33843599

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Care Management | Skills Training | Usual Care
Started | 6314 | 6312 | 6256
Completed | 6230 | 6227 | 6187
Not Completed | 84 | 85 | 69
Not completed — Disenrolled or died prior to first follow-up day - not included in outcome or adverse event counts | 84 | 85 | 69

BASELINE CHARACTERISTICS:
Population: Analysis population excludes randomized participants who died or disenrolled prior to first follow-up day
Groups:
- Total: Total of all reporting groups
Arm/Group | Care Management | Skills Training | Usual Care | Total
Number analyzed (Participants) | 6230 | 6227 | 6187 | 18644
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5254 | 5293 | 5280 | 15827
  >=65 years | 976 | 934 | 907 | 2817
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4195 | 4160 | 4188 | 12543
  Male | 2035 | 2067 | 1999 | 6101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 4723 | 4651 | 4561 | 13935
  Hispanic | 495 | 495 | 595 | 1585
  Asian, Non-Hispanic | 179 | 183 | 194 | 556
  Black, Non-Hispanic | 241 | 272 | 237 | 750
  American Indian, Non-Hispanic | 56 | 42 | 35 | 133
  Native Hawaiian or Pacific Islander | 24 | 29 | 23 | 76
  More than one race | 170 | 188 | 203 | 561
  Other or not recorded | 342 | 376 | 399 | 1117
Region of Enrollment [Number; unit: participants]
  United States | 6230 | 6227 | 6187 | 18644
Site of recruitment [Count of Participants; unit: Participants]
  Mental Health Specialty Clinic | 3071 | 3111 | 3040 | 9222
  General Medical Clinic | 3159 | 3116 | 3147 | 9422
PHQ9 item 9 score [Count of Participants; unit: Participants]
  More than half the days | 4180 | 4177 | 4141 | 12498
  Nearly every day | 2050 | 2050 | 2046 | 6146

OUTCOME MEASURES:

1. Primary Outcome: Time to Fatal or Non-fatal Suicide Attempt or Self-Harm
Description: Electronic health records and insurance claims data will be searched for any nonfatal suicide attempts or self-harm during the 18 months after randomization. Fatal suicide attempts will be identified from state mortality data.
Time Frame: 18 Months after randomization
Population: Participants were analyzed according to initial assignment, regardless of intervention participation. Follow-up time was censored at time of disenrollment from the participating health system or death due to cause other than self-harm.
Measure: Median (Inter-Quartile Range); unit: Days of follow-up time
Arm/Group | Care Management | Skills Training | Usual Care
Number analyzed (Participants) | 6230 | 6227 | 6187
Days of follow-up time | 548 [404 to 548] | 548 [398 to 548] | 548 [409 to 548]
Statistical Analysis 1: Comparison: Care Management vs Usual Care; Comparison of participants assigned to Care Management intervention to those assigned to continued Usual Care; Test type: Superiority; p = 0.61, Log Rank — A priori two-sided comparison of Care Management condition to Usual Care; A priori Bonferonni-corrected threshold for statistical significance was 0.025; Cox Proportional Hazard = 1.07, 95% CI 2-sided [0.86 to 1.33], Standard Error of Mean 0.12 — To clarify direction of comparison: relative hazard of suicide attempt among participants assigned to Care Management was 1.07 (95% CI 0.86 - 1.33) higher compared to participants assigned to Usual Care
Statistical Analysis 2: Comparison: Skills Training vs Usual Care; Comparison of Skills Training to Usual Care; Test type: Superiority — A priori two-sided comparison of Skills Training to usual care; p = 0.02, Log Rank — A priori Bonferonni-corrected threshold for statistical significance was 0.025; Cox Proportional Hazard = 1.29, 95% CI 2-sided [1.05 to 1.59], Standard Error of Mean 0.14 — To clarify direction of comparison: relative hazard of suicide attempt in participants assigned to Skills Training was 1.29 (95% CI 1.05-1.59) times higher than in those assigned to Usual Care

ADVERSE EVENTS:
Time Frame: Adverse events were ascertained for up to 18 months after randomization, censored at time of death or disenrollment from the participating health systems.
Description: Mortality was ascertained by linkage to state mortality data. Serious adverse events: Suicide attempts leading to hospitalization were ascertained from electronic health records and insurance claims data. No other adverse events were ascertained, collected, or recorded.
Arm/Group | Care Management | Skills Training | Usual Care
All-Cause Mortality (participants affected / at risk) | 133/6230 | 132/6227 | 118/6187
Serious Adverse Events (participants affected / at risk) | 71/6230 | 92/6227 | 69/6187
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Care Management (N=6230) | Skills Training (N=6227) | Usual Care (N=6187)
Self-harm leading to death or hospitalization (Psychiatric disorders) | 71 (71) | 92 (92) | 69 (69)

LIMITATIONS AND CAVEATS:
Participation in interventions was relatively low (but this reflects "real world" conditions.

Interventions could have influenced likelihood that self-harm would lead to care-seeking or be recognized and recorded by treating clinicians.

Usual care in other settings might differ from usual care in these four health systems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT02326883/Prot_SAP_000.pdf